CLINICAL TRIAL: NCT04242186
Title: Nursing Home Prevention of Injury in Dementia (NH PRIDE)
Acronym: NH PRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Duke University (Other); Brown University (Other)
Responsible Party: Principal Investigator, Sarah Berry, Associate Professor in Medicine, Hebrew SeniorLife
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-2019-21; 1R01AG062492-01 (NIH)
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Results first posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Accidental Falls/Prevention and Control
Keywords: Nursing Homes; Elderly; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nursing home residents and staff (Experimental): Nursing home residents at high risk for injurious falls, as well as nursing home staff at participating facilities
  Interventions: Other: Injury Liaison Service

INTERVENTIONS:
Other: Injury Liaison Service — The Injury Liaison Service nurse will coordinate deprescribing of fall-related medications, osteoporosis management, staff support of behavior management using video case conferencing, and shared decision making with residents and/or families.

SUMMARY:
The purpose of this study is to develop a consistent approach to prevent falls with injury in nursing home (NH) residents. A centralized Injury Liaison Service (ILS) will be developed and tested in four nursing home facilities (two in the Durham, North Carolina area and two in the Boston, Massachusetts area). The ILS will combine successful elements of a Fracture Liaison Service (FLS) and video telehealth staff education (ECHO) models with the goal of decreasing injurious falls in nursing home residents.

The ILS Program has four main components:

1. Automated identification of NH residents at high risk for falls with injury
2. Recommendations by the ILS nurse to manage medications, including deprescribing medications associated with falls and a prescription for osteoporosis medications
3. Video telehealth sessions to educate staff
4. Shared decision making with residents and/or families.

The central hypothesis of this study is that the ILS model will reduce injurious falls by changing care delivery in two areas: deprescribing psychoactive and cardiometabolic drugs to reduce falls, and increasing osteoporosis treatment to prevent injury in the setting of a fall.

Qualitative interviews will be conducted with nursing home staff to gain a better understanding of effective and non-effective injury prevention strategies. Information from these interviews will be incorporated into the study design. Outcome measures will focus on acceptability, demand, practicality, and feasibility of the program, as well as safety.

ELIGIBILITY:
Inclusion Criteria:

Facility inclusion criteria:

1. More than 80 long-stay beds
2. Within 30 miles of Boston, Massachusetts or Durham, North Carolina

Resident inclusion criteria:

1. Age ≥ 60 years
2. NH length of stay ≥ 30 days
3. Estimated 2-year risk of hip fracture ≥ 6% using FRAiL model

Provider inclusion criteria:

The NH-PRIDE intervention will target the "usual" providers including nurses, certified nursing assistants (CNAs), physicians, nurse practitioners (NPs), and physician assistants (PAs) routinely caring for NH patients. Nurses should be providing care at a NH facility for a minimum of 2 shifts most weeks. Physicians, NPs, and PAs should spend, on average a minimum of four hours weekly in nursing home care. We estimate there will be 10 providers for the qualitative interviews on injurious falls prevention, 20 providers (4 from each facility) in the televideo sessions, and 60 providers (15 per facility) to participate in the post-intervention questionnaires.

Additional eligibility criteria for providers include:

1. Worked in the facility for ≥ 90 days
2. Can communicate in English (in order to participate in interviews and questionnaires),
3. Over 21 years of age.

Proxy/resident inclusion criteria:

We will recruit 10 residents/proxies to participate in qualitative interviews on falls prevention. Residents/family must meet the following criteria:

1. Affiliated resident has lived in the facility for ≥ 30 days
2. Can communicate in English
3. Over 21 years of age
4. Able to provide informed consent to participate in the interviews

Exclusion Criteria:

Facility exclusion criteria:

1. Population not primarily English speaking
2. Evidence of institutional instability at time of recruitment

Provider exclusion criteria:

1. Does not provide routine care to NH residents (e.g., visiting hospice provider)
2. Does not speak English
3. Is less than 21 years old

Resident exclusion criteria:

1. Advanced dementia as defined by Cognitive Performance Scale (CPS) = 6
2. Life expectancy < 6 months, as indicated by Minimum Data Set (MDS) assessment
3. Living in nursing home for less than 30 days
4. Proxy has communicated wish to opt-out of study Residents will not be excluded from the study based on any specific diagnosis (e.g., congestive heart failure or schizophrenia); however, the algorithm used to make recommendations for medication management will consider individual co-morbidities.

Proxy/resident exclusion criteria for interviews:

1. Affiliated resident has lived in the facility for < 30 days
2. Cannot communicate in English
3. Less than 21 years of age
4. Unable to provide informed consent to participate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah D Berry, MD, MPH, Principal Investigator — Hebrew Rehabilitation Center; Cathleen S Colón-Emeric, MD, MHS, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Hebrew SeniorLife, Boston, Massachusetts
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Little MO, Hecker EJ, Colon-Emeric CS, Herndon L, McConnell ES, Xue TM, Berry SD. Perspectives on Deprescribing in long-term care: qualitative findings from nurses, aides, residents, and proxies. BMC Nurs. 2023 Jan 31;22(1):27. doi: 10.1186/s12912-023-01179-y. PMID 36721150
- See also: The Fracture Risk Assessment in Long term care (FRAiL) model — https://ifar-frail.hsl.harvard.edu/web/evaluation

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nursing Home Residents and Staff
Started | 140
Qualitative Interview Participants | 28
Nursing Home Residents | 46
Facility Staff Members | 66
Completed | 135
Not Completed | 5
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Groups:
- Nursing Home Residents and Staff: Nursing home residents at high risk for injurious falls, as well as nursing home staff at participating facilities. Participants included 46 nursing home residents, 28 qualitative interview participants, and 66 facility staff members.
  Injury Liaison Service: The Injury Liaison Service nurse will coordinate deprescribing of fall-related medications, osteoporosis management, staff support of behavior management using video case conferencing, and shared decision making with residents and/or families.
Arm/Group | Nursing Home Residents and Staff
Number analyzed (Participants) | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 94
  >=65 years | 46
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Continuous age data are included only for nursing home residents. Continuous age data were not collected from interview participants and staff members.
  years
    number analyzed (Participants) | 46
    (all) | 88 [81 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 140

OUTCOME MEASURES:

1. Primary Outcome: Number of High-risk Residents According to the FRAiL Model
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Groups:
- Nursing Home Residents: Nursing home residents at high risk for injurious falls
Arm/Group | Nursing Home Residents
Number analyzed (Participants) | 46
Participants | 46

2. Primary Outcome: Number of High-risk Residents With One or More Deprescribing Recommendations
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nursing Home Residents
Number analyzed (Participants) | 46
Participants | 36

3. Primary Outcome: Number of Residents Whose Provider Accepted One or More Deprescribing Recommendations
Time Frame: 4 months
Population: 36 participants had one or more deprescribing recommendations
Measure: Count of Participants; unit: Participants
Arm/Group | Nursing Home Residents
Number analyzed (Participants) | 36
Participants | 21

4. Primary Outcome: Number of Residents Who Accepted One or More Deprescribing Recommendations
Time Frame: 4 months
Population: 21 residents had deprescribing recommendations accepted by their provider
Measure: Count of Participants; unit: Participants
Arm/Group | Nursing Home Residents
Number analyzed (Participants) | 21
Participants | 21

5. Primary Outcome: Number of High-risk Residents With a Recommendation for Osteoporosis Treatment
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nursing Home Residents
Number analyzed (Participants) | 46
Participants | 20

6. Primary Outcome: Number of Residents Whose Provider Accepted Osteoporosis Treatment Recommendations
Time Frame: 4 months
Population: 20 participants had a recommendation for osteoporosis treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nursing Home Residents
Number analyzed (Participants) | 20
Participants | 10

7. Primary Outcome: Number of Residents Who Accepted Osteoporosis Treatment Recommendations
Time Frame: 4 months
Population: 10 residents had osteoporosis treatment recommendations accepted by their provider
Measure: Count of Participants; unit: Participants
Arm/Group | Nursing Home Residents
Number analyzed (Participants) | 10
Participants | 10

8. Primary Outcome: Attrition of Eligible Residents From the NH Facility Due to Transfer, Discharge to Community, or Death
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nursing Home Residents
Number analyzed (Participants) | 46
Participants | 6

9. Primary Outcome: Proportion of Staff Members Who Indicated They Were Satisfied or Very Satisfied With the ILS on a Post-intervention Survey
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Nursing Home Staff: Staff who participated in the program and completed a satisfaction survey
Arm/Group | Nursing Home Staff
Number analyzed (Participants) | 21
Participants | 17

10. Primary Outcome: Number of Staff Members Who Attended One or More ECHO Sessions
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nursing Home Staff
Number analyzed (Participants) | 21
Participants | 21

11. Secondary Outcome: Average Number of Deprescribing Recommendations That Were Made for Each Resident
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: number of recommendations
Arm/Group | Nursing Home Residents
Number analyzed (Participants) | 46
number of recommendations | 2.2 (1.3)

12. Secondary Outcome: Average Number of Adverse Drug Events
Description: 1. Escalating behaviors, worsening depression, or functional decline following psychoactive medication deprescribing
  2. Unplanned medical visits for hypertension, tachycardia, or hyperglycemia following cardiometabolic deprescribing
  3. New gastroesophageal reflux disease or esophagitis following bisphosphonate prescription
  Adverse drug events were analyzed in residents who had one or more medications deprescribed (n=21).
Time Frame: 4 months
Population: Adverse drug events were analyzed in residents who had one or more medications deprescribed (n=21).
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Nursing Home Residents
Number analyzed (Participants) | 21
number of events | 0.05 (0.22)

13. Secondary Outcome: Number of Injurious Falls
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: number of injurious falls
Arm/Group | Nursing Home Residents
Number analyzed (Participants) | 46
number of injurious falls | 0.07 (0.25)

ADVERSE EVENTS:
Time Frame: 4 months
Description: We used the clinicaltrials.gov definitions of adverse events. All-Cause Mortality, Serious Adverse Events and Other Adverse Events were not monitored/assessed in facility staff. They were only assessed in nursing home residents at high risk for falls (n=46).
Groups:
- Nursing Home Residents: Adverse events were monitored in nursing home residents at high risk for injurious falls (n=46)
Arm/Group | Nursing Home Residents
All-Cause Mortality (participants affected / at risk) | 5/46
Serious Adverse Events (participants affected / at risk) | 9/46
Other Adverse Events (participants affected / at risk) | 1/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nursing Home Residents (N=46)
Intraventricular hemorrhage following a fall and resulting in death (Infections and infestations) | 1 (1)
Advanced dementia resulting in death (Nervous system disorders) | 3 (3)
Suspected cardiac event resulting in death (Cardiac disorders) | 1 (1)
Urosepsis resulting in hospitalization (Infections and infestations) | 2 (2)
Agitation and aggression resulting in hospitalization (Nervous system disorders) | 1 (1)
Acute colitis resulting in hospitalization (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nursing Home Residents (N=46)
Adverse drug withdrawal event (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT04242186/Prot_SAP_000.pdf
  • Informed Consent Form: Proxy ICF (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT04242186/ICF_001.pdf
  • Informed Consent Form: Provider ICF (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT04242186/ICF_002.pdf